CLINICAL TRIAL: NCT00623584
Title: In Vitro and Clinical Comparison of Corneal Grafts Cultured in Serum Free Medium or Standard Serum Supplemented Medium in Patients With Degeneration of the Corneal Endothelium
Brief Title: Comparison of Corneal Grafts Cultured in Serum-free Versus Corneal Grafts Cultured in Serum Supplemented Culture Media
Acronym: SFM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Klinikum Chemnitz gGmbH (Other)
Collaborators: German Research Foundation (Other); KKS Netzwerk (Network)
Responsible Party: Prof. Dr. med. Katrin Engelmann, Eye Clinic Chemnitz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKC001SFM08
Record Dates: First submitted 2008-02-13; First posted 2008-02-26 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Fuch's Endothelial Dystrophy; Pseudophakic Bullous Keratopathy
Keywords: penetrating keratoplasty; corneal transplantation; corneal grafting; corneal grafts; culture media; corneal culturing; in vitro culturing
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy | interventions — Corneal Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients in this arm randomly receive a corneal graft cultured in a serum free culture medium
  Interventions: Procedure: Corneal transplantation
- 2 (Active Comparator): Patients in this arm randomly receive a corneal graft cultured in a serum supplemented culture medium
  Interventions: Procedure: Corneal transplantation

INTERVENTIONS:
Procedure: Corneal transplantation — Full thickness penetrating keratoplasty
  Arms: 1
Procedure: Corneal transplantation — Full thickness penetrating keratoplasty
  Arms: 2

SUMMARY:
The goal of this clinical trial is to compare the quality of corneal grafts cultured in a serum-free culture medium with a defined composition versus corneal grafts cultured in a standard serum supplemented culture medium transplanted in patients with decompensated corneal dystrophy

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to test the equivalence of the quality of the corneal grafts cultured under serum free conditions to corneal grafts cultured in the Minimal Essential Medium supplemented with 2% fetal calf serum, based on a parallel comparison of the endothelial cell density of paired corneal grafts deriving from single donors at different time points before and after the grafting procedure. In addition, the safety of the clinical use of corneal grafts cultured in both media will be determined. The graft survival rate during the follow-up period will be quantified in regard to immune mediated graft rejection and non-immune mediated graft failure, as well as the incidence of corneal edema, corneal opacities and corneal neovascularisation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 50 and 85 years of age
* Clinically proven Fuchs corneal dystrophy or secondary decompensation the corneal endothelium (e. g. after surgical intervention in the anterior segment of the eye)
* Patient informed consent

Exclusion Criteria:

* Previous penetrating keratoplasty
* Corneal neovascularisation
* Pathologic changes in the anterior segment of the eye (anterior / posterior synechiae, uveitis)
* Glaucoma
* Aphakia
* Infectious diseases of the cornea
* Neurodermitis
* Participation of the patient in another clinical trial within the last four weeks that precede the recruitment
* The patient is unlikely to comply with the requirements of the protocol
* Previous or current abuse of medications, narcotics or alcohol
* Pregnancy

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the endothelial cell density of the corneal grafts prior to and after the transplantation procedure | The measurment will be performed prior to and 1, 4, 12, 24, 36, 48 and 60 months after the transplantation

SECONDARY OUTCOMES:
Secondary study outcomes are immune mediated graft rejection, non-immune mediated graft failure, as well as the incidence of corneal edema, corneal opacities and corneal neovascularisation. | 1,4,12, 24, 36, 48 and 60 month after the transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Engelmann, MD, Principal Investigator — Klinikum Chemnitz GmbH
Locations (2):
- Germany (2):
  - Augenklinik, Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Universitäts Augenklinik, Halle, Saxony-Anhalt

REFERENCES:
- [Background] Hempel B, Bednarz J, Engelmann K. Use of a serum-free medium for long-term storage of human corneas. Influence on endothelial cell density and corneal metabolism. Graefes Arch Clin Exp Ophthalmol. 2001 Oct;239(10):801-5. doi: 10.1007/s004170100364. PMID 11760044
- [Background] Bednarz J, Doubilei V, Wollnik PC, Engelmann K. Effect of three different media on serum free culture of donor corneas and isolated human corneal endothelial cells. Br J Ophthalmol. 2001 Dec;85(12):1416-20. doi: 10.1136/bjo.85.12.1416. PMID 11734511
- [Background] Uphoff J, Bednarz J, Engelmann K. [Follow-up of endothelial cell density after perforating keratoplasty. Effect of donor and recipient-related factors]. Ophthalmologe. 2001 Jun;98(6):550-4. doi: 10.1007/s003470170117. German. PMID 11450479
- [Background] Moller-Pedersen T, Hartmann U, Moller HJ, Ehlers N, Engelmann K. Evaluation of potential organ culture media for eye banking using human donor corneas. Br J Ophthalmol. 2001 Sep;85(9):1075-9. doi: 10.1136/bjo.85.9.1075. PMID 11520760
- [Background] Moller-Pedersen T, Hartmann U, Ehlers N, Engelmann K. Evaluation of potential organ culture media for eye banking using a human corneal endothelial cell growth assay. Graefes Arch Clin Exp Ophthalmol. 2001 Oct;239(10):778-82. doi: 10.1007/s004170100354. PMID 11760040